CLINICAL TRIAL: NCT00345072
Title: A Menopause Interactive Decision Aid System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: R01HS013329-02 (AHRQ)
Record Dates: First submitted 2006-06-26; First posted 2006-06-27 (Estimated); Last update posted 2006-06-27 (Estimated); Status verified 2006-06

CONDITIONS: Menopause
Keywords: Menopause; Decision aids; Internet; Hormone Replacement Therapy; Breast Cancer; Cardiovascular Disease; Osteoporosis
MeSH Terms: conditions — Breast Neoplasms; Cardiovascular Diseases; Osteoporosis

INTERVENTIONS:
Device: Web-based decision aid system

SUMMARY:
The purpose of this study is to develop and test a web-based system intended to help women going through menopause make more informed choices regarding menopause treatments. The system will do this by giving women personalized feedback on the risks and benefits of these treatments.

DETAILED DESCRIPTION:
Most women are not satisfied with the counseling they receive about menopause. To improve menopause counseling and help menopausal women more actively participate in the decision making process, we have developed a novel prototype web-based decision aid. Our immediate goal is to develop this prototype technology into a comprehensive Menopause Interactive Decision Aid System (MIDAS) that provides personalized feedback about menopausal symptoms, risks for common conditions, and the effects of different treatment options on the short- and long-term consequences of menopause.

Our main study hypotheses are that MIDAS can: 1) lead to better decisions and improve the quality of menopausal counseling; 2) improve compliance with a chosen menopausal plan; and 3) reduce medical errors associated with the use of menopausal therapies.

We propose a 2-phase study conducted over 3 years. Phase I will transform the prototype application into a comprehensive MIDAS, completing its content and risk assessment instruments, and exploring its optimal design. This will be accomplished through conduct of focus groups and usability tests. Phase II will formally evaluate the impact of MIDAS in a randomized, controlled, multi-center clinical trial involving diverse patient populations and clinician settings. We will measure the impact of MIDAS on the decision-making process as well as its effect on providers and outcome measures related to menopause, including compliance, quality of life, and medical errors related to menopausal therapy. Analyses will evaluate the extent to which the impact of MIDAS on these outcomes varies according to patient, practice, and physician characteristics.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Between 45 and 65 years of age
* Patient at participating clinics
* Experience menopausal symptoms or being 6 months or more past last menstrual period
* Have an upcoming appointment for menopausal counseling or annual physical exam (only applicable for clinical trial participants)

Exclusion Criteria:

* Inability to give informed consent
* Dementia
* Age over 65 years
* Pre-existing terminal illness that limits life expectancy to less than 2 years
* History of breast cancer or cardiovascular disease

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 296
Dates: Start 2003-07

PRIMARY OUTCOMES:
Decisional conflict
Knowledge of the benefits, risks and side effects of menopausal treatments
Risk perception for breast cancer, CHD, and hip fracture
Patient-physician communication
Satisfaction with decision
Anxiety
Depression
Quality of menopausal counseling
Adherence to medication and lifestyle changes
Health-related quality of life
Menopause-specific quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Nananda F Col, MD, MPH, MPP, Principal Investigator — Rhode Island Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Rhode Island Hospital, Providence, Rhode Island